CLINICAL TRIAL: NCT04655443
Title: Risk Factors That Contribute to the Maintenance of Sinus Rhythm: A Prospective Study to Create a Prediction Model for Atrial Fibrillation Patients to Maintain Sinus Rhythm.
Brief Title: Risk Factors That Contribute to the Maintenance of Sinus Rhythm
Acronym: Afib
Status: Terminated | Type: Observational
Why Stopped: due to COVID-19
Sponsor: Danbury Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 17-601
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Patients will be scheduled for an electrocardiogram thirty days after their electrical cardioversion. Based on the electrocardiogram result, patients that maintained sinus rhythm will be assigned to "Control".
  Interventions: Other: Standard Care
- Afib Group: Patients will be scheduled for an electrocardiogram thirty days after their electrical cardioversion. Based on the electrocardiogram result, patients that developed persistent atrial fibrillation will be assigned to "Afib".
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Standard Care — Standard cardiovascular care

SUMMARY:
This is a prospective clinical research study. The objective of this study is to evaluate if clinical risk factors as well as structural features on echocardiography affect the maintenance of sinus rhythm after electrical cardioversion at 30 days. The investigators anticipate 140 patients to be enrolled in the study.

DETAILED DESCRIPTION:
Atrial fibrillation is the most commonly diagnosed arrhythmia in the United States. A systematic review of worldwide population-based studies estimated that approximately 33 million people were diagnosed with atrial fibrillation in 2010. The prevalence of atrial fibrillation in the United States increases with advancing age. Approximately 1% of patients with atrial fibrillation are under 60 years of age whereas more than one-third are over 80 years of age.

Although atrial fibrillation is commonly diagnosed and continues to have increased incidence in the country, patients continue to be admitted to the hospital for worsening symptoms of chest pain, shortness of breath, and palpitations. Long-term complications of atrial fibrillation include cardiomyopathy, cerebrovascular events, thromboembolic events, and death.

Many medications have been established to convert patients from atrial fibrillation to normal sinus rhythm; however procedures of cardioversion and ablation have also proven to be effective. A study, the AFFIRM trial, published in the New England Journal of Medicine in 2002 discussed the benefit of converting patients to sinus rhythm versus keeping patients in atrial fibrillation, however making sure their heart rates were well-controlled. This study did not demonstrate a significant difference in death, ischemic stroke, or major bleeding in both treatment arms suggesting there is no benefit of converting patients from atrial fibrillation to normal sinus rhythm. However, with increasing health costs occurring around the country, every effort should be made to help improve patient symptoms and avoid unnecessary hospitalizations. A study published in the Journal of American College of Cardiology in 2004, "Effect of rate or rhythm control on quality of life in persistent atrial fibrillation: Results from the Rate Control Versus Electrical Cardioversion (RACE) study," concluded that the quality of life was impaired in patients with atrial fibrillation. Another study published in 2012, "Economic Burden of Atrial Fibrillation: Implications for Intervention," reported total costs of atrial fibrillation care in the United States to be estimated to be $6.65 billion per year.

Our study is designed to look at patients with atrial fibrillation who underwent electrical cardioversion to restore sinus rhythm and create a prediction model to identify specific risk factors, which may contribute to persistent atrial fibrillation.

Prediction models have been established in regards to maintaining sinus rhythm, including the Hatch Score, which examined risk factors of hypertension, history of TIA or stroke, chronic obstructive pulmonary disease, and heart failure that predisposed patients to persistent atrial fibrillation. Another score established was the LADS score, which observed risk factors of left atrial diameter, age, history of stroke, and smoking status as predictors of persistent atrial fibrillation. The purpose of our study is to create a new prediction model using clinical and echocardiographic parameters to determine if these factors will predict persistent atrial fibrillation after electrical cardioversion. Transesophageal echocardiographic parameters include imaging of the left atrial appendage (LAA) and calculating the LAA ejection fraction (LAAEF) by 3D or biplane Simpson method (based on image quality), and using pulse-wave Doppler to calculate the LAA exit velocity and S/D ratio across the pulmonic vein. Transthoracic echocardiographic parameters include estimated pulmonary arterial pressure (PASP) using tricuspid regurgitation (TR) jet velocity, left atrial volume index (LAVi), left ventricular (LV) size, LV hypertrophy (LVH) and left ventricular ejection fraction (LVEF).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Documented atrial fibrillation by electrocardiogram (ECG)
* Patients undergoing electrical cardioversion for atrial fibrillation
* Patients with a baseline transthoracic echocardiography within 1 month prior to the cardioversion

Exclusion Criteria:

* Patients who did not convert to normal sinus rhythm after electrical cardioversion
* Patients who are found to have a LAA thrombus on TEE
* Patients who do not have a follow up ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing electrical cardioversion for atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Transthoracic Echocardiography and Transesophageal Echocardiography findings | 30 days post electrical cardioversion
  Left ventricular ejection fraction, left ventricular size, left ventricular hypertrophy, left atrial volume index, mitral valve early diastolic inflow velocity E, mitral valve tissue Doppler velocity e', E/e' ratio and pulmonary arterial pressure will be collected from transthoracic echocardiography findings in medical record. Left atrial size, left atrial appendage ejection fraction, left atrial appendage exit velocity, pulmonary venous flow with S/D ratio, and presence of spontaneous echo contrast will be collected from transesophageal echocardiography findings in medical record. Transthoracic Echocardiography and Transesophageal Echocardiography findings between participants that maintained sinus rhythm and participants that developed persistent atrial fibrillation will be compared to create a prediction model to identify specific risk factors, which may contribute to persistent atrial fibrillation.

SECONDARY OUTCOMES:
Clinical risk factors | 30 days post electrical cardioversion
  History of stroke/transient ischemic attack, hypertension, diabetes mellitus, congestive heart failure, coronary artery disease, pulmonary hypertension, chronic obstructive pulmonary disease, sleep apnea, hyperthyroidism, obesity, tobacco use, alcohol use, and home medications will be collected from medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Galin, MD, Principal Investigator — Danbury Hospital, Nuvance Health
Locations (1):
- Danbury Hospital, Danbury, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):e199-267. doi: 10.1161/CIR.0000000000000041. Epub 2014 Mar 28. No abstract available. PMID 24682347
- [Result] Vlachos K, Letsas KP, Korantzopoulos P, Liu T, Georgopoulos S, Bakalakos A, Karamichalakis N, Xydonas S, Efremidis M, Sideris A. Prediction of atrial fibrillation development and progression: Current perspectives. World J Cardiol. 2016 Mar 26;8(3):267-76. doi: 10.4330/wjc.v8.i3.267. PMID 27022458
- [Result] Wyse DG, Waldo AL, DiMarco JP, Domanski MJ, Rosenberg Y, Schron EB, Kellen JC, Greene HL, Mickel MC, Dalquist JE, Corley SD; Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) Investigators. A comparison of rate control and rhythm control in patients with atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1825-33. doi: 10.1056/NEJMoa021328. PMID 12466506
- [Result] Kim MH, Johnston SS, Chu BC, Dalal MR, Schulman KL. Estimation of total incremental health care costs in patients with atrial fibrillation in the United States. Circ Cardiovasc Qual Outcomes. 2011 May;4(3):313-20. doi: 10.1161/CIRCOUTCOMES.110.958165. Epub 2011 May 3. PMID 21540439
- [Result] Gilbert KA, Hogarth AJ, MacDonald W, Lewis NT, Tan LB, Tayebjee MH. Restoration of sinus rhythm results in early and late improvements in the functional reserve of the heart following direct current cardioversion of persistent AF: FRESH-AF. Int J Cardiol. 2015 Nov 15;199:121-5. doi: 10.1016/j.ijcard.2015.07.020. Epub 2015 Jul 11. PMID 26188832
- [Result] Ecker V, Knoery C, Rushworth G, Rudd I, Ortner A, Begley D, Leslie SJ. A review of factors associated with maintenance of sinus rhythm after elective electrical cardioversion for atrial fibrillation. Clin Cardiol. 2018 Jun;41(6):862-870. doi: 10.1002/clc.22931. Epub 2018 Jun 7. PMID 29878481
- [Result] Malik S, Hicks WJ, Schultz L, Penstone P, Gardner J, Katramados AM, Russman AN, Mitsias P, Silver B. Development of a scoring system for atrial fibrillation in acute stroke and transient ischemic attack patients: the LADS scoring system. J Neurol Sci. 2011 Feb 15;301(1-2):27-30. doi: 10.1016/j.jns.2010.11.011. Epub 2010 Dec 4. PMID 21130468
- [Result] European Heart Rhythm Association; Heart Rhythm Society; Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Zamorano JL; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines; Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation. ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation). J Am Coll Cardiol. 2006 Aug 15;48(4):854-906. doi: 10.1016/j.jacc.2006.07.009. No abstract available. PMID 16904574
- [Result] Akdemir B, Altekin RE, Kucuk M, Yanikoglu A, Karakas MS, Aktas A, Demir I, Ermis C. The significance of the left atrial volume index in cardioversion success and its relationship with recurrence in patients with non-valvular atrial fibrillation subjected to electrical cardioversion: a study on diagnostic accuracy. Anadolu Kardiyol Derg. 2013 Feb;13(1):18-25. doi: 10.5152/akd.2013.003. Epub 2012 Oct 12. PMID 23070632
- [Result] Antonielli E, Pizzuti A, Palinkas A, Tanga M, Gruber N, Michelassi C, Varga A, Bonzano A, Gandolfo N, Halmai L, Bassignana A, Imran MB, Delnevo F, Csanady M, Picano E. Clinical value of left atrial appendage flow for prediction of long-term sinus rhythm maintenance in patients with nonvalvular atrial fibrillation. J Am Coll Cardiol. 2002 May 1;39(9):1443-9. doi: 10.1016/s0735-1097(02)01800-4. PMID 11985905